CLINICAL TRIAL: NCT06960564
Title: Investigation of the Effect of Hyaluronic Acid Injection on Tnf-Alpha and IL-1beta at DNA-Protein Level in Knee Osteoarthritis Patients and Comparison With Clinical Parameters: A Randomised Controlled Trial
Brief Title: The Effect of Hyaluronic Acid Injection on TNF-Alpha and IL-1β in Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: Istanbul University Research Fund (Unknown)
Responsible Party: Principal Investigator, Dicle Rotinda Ozdas Sevgin, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-68869993-511.06.01.01-159494
Record Dates: First submitted 2025-04-28; First posted 2025-05-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-06

CONDITIONS: Knee Osteoarthritis; Hyaluronic Acid
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra-articular hyaluronic acid injection group (Active Comparator)
  Interventions: Device: Hyaluronic Acid injections
- Intra-articular saline injection group (Placebo Comparator)
  Interventions: Other: Saline -- placebo comparator

INTERVENTIONS:
Device: Hyaluronic Acid injections — Intra-articular hyaluronic acid will be administered to 30 selected patients. Blood and synovial fluid samples will be collected before HA injection and 1 week after 3 sessions of HA injection with one week interval. Home exercise programme will be given.
  Arms: Intra-articular hyaluronic acid injection group
Other: Saline -- placebo comparator — Intra-articular saline (SF) will be administered to 20 selected patients. Blood and synovial fluid samples will be collected before and 1 week after 3 session of salin injection with one week interval. Home exercise programme will be given.
  Arms: Intra-articular saline injection group

SUMMARY:
In this study, the effect of intra-articular HA injection therapy on pre- and post-treatment TNF-alpha and IL-1beta levels and methylation changes in blood and synovial fluid in patients with knee osteoarthritis will be determined and compared with the placebo group. In addition, the effects of HA injection on pain, functional status and quality of life will be evaluated and these effects will be related to changes in TNF-alpha and IL-1-beta.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of knee osteoarthritis according to ACR (American College of Rheumatology) criteria
* Knee pain for more than 3 months
* Presence of knee pain resistant to conservative treatment for at least 3 months
* To be between the ages of 45-75
* Kellgren-Lawrence stage 2-3 gonarthrosis detected in the available knee direct radiographs of the patients

Exclusion Criteria:

* Patients with KL stage 1 and 4 OA
* Systematic diseases (severe cardiovascular disease, severe renal failure, severe hepatic failure, uncontrolled diabetes, cancer, immunosuppression, haematological diseases, systemic bone diseases)
* Bleeding tendency (acquired or inherited) [lNR>2 in a patient on Coumadin],
* Infection (systemic or local)
* Secondary knee osteoarthritis (inflammatory joint disease, post-traumatic, post-infectious, etc.)
* Major knee trauma within the last 1 year
* BMI >40
* History of total knee or hip arthroplasty within 1 year
* Pregnancy
* History of intra-articular injection within the last 6 months
* Patients with Hb less than 11 g/dl and Plt less than 150.000
* Presence of allergy to hyaluronic acid products

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-03-29 (Estimated)

PRIMARY OUTCOMES:
Blood and synovial fluid TNF-alpha levels | Assessments will be made before and 1 week after treatment
Blood and synovial fluid IL-1beta levels | Assessments will be made before and 1 week after treatment
Blood and synovial fluid TNF-alpha methylation changes | Assessments will be made before and 1 week after treatment
Blood and synovial fluid IL-1beta methylation changes | Assessments will be made before and 1 week after treatment

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS)-pain (activity, rest, night) | Evaluations will be performed before and 1 month, 3 months and 6 months after treatment
  minimum value : 0 maximum value :10 Higher scores mean worse outcome.
The Western Ontario and McMaster Universities Arthritis Index (WOMAC)- (pain, stiffness, physical function, total score) | Evaluations will be performed before and 1 month, 3 months and 6 months after treatment
  Minimum value: 0 maximum value : 96 Higher scores mean worse outcome
Lequesne Index (pain or discomfort, walking distance, GYA) | Evaluations will be performed before and 1 month, 3 months and 6 months after treatment
  Minimum value : 0 maximum value: 24 higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided